CLINICAL TRIAL: NCT03651245
Title: European Alpha-Mannosidosis Participant: An International, Multicenter, Epidemiological Protocol
Brief Title: European Alpha-Mannosidosis Participant
Acronym: EUMAP
Status: Terminated | Type: Observational
Why Stopped: we will update quickly
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: EUMAP-2018
Record Dates: First submitted 2018-08-24; First posted 2018-08-29 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Immunodeficiency; Skeletal Abnormalities; Deafness; Mental Retardation; Gingival Hypertrophy; Facial Dysmorphism
Keywords: Alpha-Mannosidosis disease; prevalence
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Deafness; Intellectual Disability; Gingival Hypertrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample applied on the Dry Blood Spot (DBS) Filtercard (Centocard®)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with suspicion for Alpha-Mannosidosis: Participants with suspicion for Alpha-Mannosidosis based on their clinical symptoms aged from 2 months to 18 years

SUMMARY:
International, multicenter, observational, longitudinal monitoring study to investigate the prevalence of Alpha-Mannosidosis in participants at risk for Alpha-Mannosidosis.

DETAILED DESCRIPTION:
Alpha-Mannosidosis is a lysosomal storage disorder of the Glycoprotein family of diseases and is closely related to Mucopolysaccharidoses.It is a rare inherited disorder that causes problems in many organs and tissues of the body. Affected individuals may have intellectual disability, distinctive facial features, and skeletal abnormalities. Characteristic facial features can include a large head, prominent forehead, low hairline, rounded eyebrows, large ears, flattened bridge of the nose, protruding jaw, widely spaced teeth, overgrown gums, and large tongue. The skeletal abnormalities that can occur in this disorder include reduced bone density (osteopenia), thickening of the bones at the top of the skull (calvaria), deformations of the bones in the spine (vertebrae), bowed legs or knock knees, and deterioration of the bones and joints.

Affected individuals may also experience difficulty in coordinating movements (ataxia); muscle weakness (myopathy); delay in developing motor skills such as sitting and walking; speech impairments; increased risk of infections; enlargement of the liver and spleen (hepatosplenomegaly); a buildup of fluid in the brain (hydrocephalus); hearing loss; and a clouding of the lens of the eye (cataract).

Alpha-Mannosidosis is estimated to occur in approximately 1 in 500,000 people worldwide. Mutations in the MAN2B1 gene cause Alpha-Mannosidosis. This gene provides instructions for making the enzyme alpha-mannosidase. Mutations in the MAN2B1 gene interfere with the ability of the alpha-mannosidase enzyme to perform its role in breaking down mannose-containing oligosaccharides. These oligosaccharides accumulate in the lysosomes and cause cells to malfunction and eventually die. Tissues and organs are damaged by the abnormal accumulation of oligosaccharides and the resulting cell death, leading to the characteristic features of Alpha-Mannosidosis.

Modern methods, as DBS based mass-spectrometry give a great opportunity to

* Simplify the diagnostic process
* Simplify the logistics
* Increases stability and reproducibility
* Characterize specific metabolic alterations in the blood of affected patients that allow diagnosing the disease earlier, with a higher sensitivity and specificity.

A more specific diagnosis that permits earlier detection of the disease, as well as assessment of the disease activity and progression, would also permit improved chances for earlier treatment of those patients suffering from the disease.

It is the goal of this international, multicentre, epidemiological study to explore and analyse the prevalence of Alpha-Mannosidosis disease in a cohort of 1.000 patients with a suspicion of Alpha-Mannosidosis disease, based on the patient's clinical symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent is obtained from the participant's parent/legal guardian
* The participant is aged between 2 months and 18 years of age
* The participant has a family history of Alpha-Mannosidosis or is at risk for Alpha-Mannosidosis according to one or more of the following symptoms: recurrent infections, skeletal abnormalities, hearing impairment-deafness, progressive neurological symptoms, impairment of mental functions, gingival hypertrophy, dysmorphic facial features, motoric disturbances of no obvious etiology

Exclusion Criteria:

* Informed consent is not provided by the partici-pant's parent/legal guardian
* The participant is younger than 2 months or older than 18 years
* The participant has no family history of Alpha-Mannosidosis and is not at risk for Alpha-Mannosidosis (represents none of the following symptoms): recurrent infections, skeletal abnormalities, hearing impairment-deafness, progressive neurological symptoms, impairment of mental functions, gingival hypertrophy, dysmorphic facial features, motoric disturbances of no obvious etiology

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants at risk for Alpha-Mannosidosis
Sampling Method: Probability Sample
Enrollment: 667 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Epidemiological analysis of the prevalence of Alpha-Mannosidosis disease in a cohort of patients with suspicion for Alpha-Mannosidosis, based on their clinical symptoms. | 3 years
  Number of identified Alpha-Mannosidosis patients, showing a mutation/pathogenic variant in the MAN2B1-Gene, within a cohort of 1000 suspected cases using respective patient's dry-blood sample for confirmatory genetic testing (NGS-based sequencing of MAN2B1-gene)

SECONDARY OUTCOMES:
Establishment of biomarker/s in MAN2B1 positive cohort. | 3 years
  Alpha-Mannosidosis-positive samples will be validated for the identification of potential biomarkers (based on MS/MS-Tandem spectroscopy) and compared with the merged control samples in order establish a disease-specific biomarker.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof. Dr., Study Chair — CENTOGENE GmbH
Locations (19):
- Germany (17):
  - Uniklinik RWTH Aachen Klinik für Kinder- und Jugendmedizin, Aachen
  - Charité - Universitätsmedizin Berlin, Leitung Sozialpädiatrisches Zentrum, Klinik für Pädiatrie m.S. Neurologie, Berlin
  - Carl-Thiem-Klinikum Cottbus GmbH, Klinik für Kinder und Jugendmedizin, Cottbus
  - Universitätsklinikum Essen, Klinik für Hals-Nasen und Ohrenheilkunde, Essen
  - Universitätsklinikum Gießen, Zentrum für Kinderheilkunde und Jugendmedizin, Abteilung für Kinderneurologie, Sozialpädiatrie und Epileptologie, Giessen
  - Universitätsklinikum Halle Universitätsklinik und Poliklinik für Pädiatrie I, Halle
  - UKE - Universitätsklinikum Hamburg-Eppendorf Klinik und Poliklinik für Hals-, Nasen- und Ohrenheilkunde, Hamburg
  - Evangelisches Krankenhaus Hamm, Klinik für Kinder-und Jugendmedizin, Hamm
  - Medizinische Hochschule Hannover, Deutsches HörZentrum Hannover, Hanover
  - Universitätsklinikum Jena, Klinik für Hals-, Nasen- und Ohrenheilkunde, Jena
  - Universitätsklinikum Jena, Klinik für Neuropädiatrie, Jena
  - UNIVERSITÄTSKLINIKUM LEIPZIG AöR, Klinik und Poliklinik für Hals-, Nasen-, Ohrenheilkunde, Leipzig
  - Sozialpädiatrisches Zentrum der HTZ Neuwied gGmbH, Neuwied
  - Evangelisches Krankenhaus Oberhausen, Sozialpädiatrisches Zentrum, Oberhausen
  - Elblandkliniken Stiftung & Co. KG - Elblandklinkum Riesa Sozialpädiatrisches Zentrum und Frühförderstelle, Riesa
  - Klinik für Kinder-und Jungendmedizin des Universitätsklinikums Ulm, Ulm
  - Zentrum für Kinder und Jugendliche Sozialpädiatrisches Zentrum (SPZ) im Marien-Hospital, Wesel
- Switzerland (2):
  - HNO-Universitätsklinik, Universitätsspital Basel, Basel
  - Inselspital Bern Universitätsklinik für Neurologie, Bern

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CENTOGENE is a rare disease company focused on transforming clinical, genetic, and biochemical data into medical solutions for patients — https://www.centogene.com/